CLINICAL TRIAL: NCT07101250
Title: Preoperative Acetazolamide for Improved Pain Control Following Laparoscopic Hysterectomy
Brief Title: Preoperative Acetazolamide
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2310736
Record Dates: First submitted 2025-07-25; First posted 2025-08-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Post Operative Pain; Laparoscopic Hysterectomy; Referred Pain
Keywords: shoulder pain; laparoscopic; analgesia
MeSH Terms: conditions — Pain, Postoperative; Pain, Referred; Shoulder Pain; Agnosia | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, controlled trial
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Drug (Active Comparator): Acetazolamide 500mg ER
  Interventions: Drug: Acetazolamide 500 MG Extended Release Oral Capsule
- Placebo (Active Comparator): Inactive Placebo Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide 500 MG Extended Release Oral Capsule — Active Drug
  Other Names: Diamox
  Arms: Active Drug
Drug: Placebo — Inactive Drug
  Arms: Placebo

SUMMARY:
The goal of this randomized study looks at whether giving patients a medicine called acetazolamide (also called Diamox) before they have laparoscopic hysterectomy may decrease postoperative pain. Researchers will compare acetazolamide to a placebo or inactive drug, to see if acetazolamide helps the pain that may occur after surgery from the gas used in the abdomen during the laparoscopic procedure. Patients will be asked to rate their pain before surgery and after surgery through 24 hours.

DETAILED DESCRIPTION:
Pain control following surgery is integral to surgical success, allowing faster recovery and return to function and increasing patient satisfaction. Minimally invasive surgery, such as laparoscopy, is becoming increasingly common as it involves smaller incisions and theoretically less discomfort. However, in order to perform laparoscopy, one must insufflate the abdomen with gas in order to create space in which to operate. The most commonly used gas today is carbon dioxide, as it is highly soluble and reduces the risk of air embolism compared to room air if absorbed. A consequence of using carbon dioxide is that it is converted to carbonic acid that can be irritating to the peritoneum and specifically the diaphragm, causing referred pain to the right subscapular (shoulder) region. Multiple strategies have been undertaken to help reduce this discomfort, one of which is using acetazolamide (a carbonic anhydrase inhibitor) to help reduce peritoneal acidification. Multiple studies have demonstrated an improvement in shoulder pain following preoperative administration in laparoscopic cholecystectomy, but studies evaluating use in pelvic surgery have had mixed results. The goal of this study is to add to this understanding and determine if acetazolamide is a useful adjunct to current pain control methods in laparoscopic gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Ages 21-65
* undergoing total laparoscopic hysterectomy (TLH) for benign indications with or without bilateral salpingoophorectomy
* undergoing total laparoscopic hysterectomy (TLH) for benign indications with or without cystoscopy

Exclusion Criteria:

* Allergy to acetazolamide or sulfonamides
* Known electrolyte disturbances
* Pregnancy
* Kidney failure or creatinine >1.5
* Diuretic or lithium use
* Chronic obstructive pulmonary disease (COPD) or other lung disease
* Central nervous system disorders
* Liver disease
* Glaucoma
* Preoperative or chronic opioid use
* Diagnosis of fibromyalgia
* Preoperative shoulder pain
* Conversion to laparotomy
* Intraoperative bladder or bowel injury
* Inability to understand or utilize visual analog scale
* Undergoing concurrent reconstructive procedures

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study of female surgery
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal/pelvic pain and right subscapular pain rated on a VAS at five perioperative points | From before procedure to 24 hours post procedure
  Baseline score at preoperative time point and 4 time points post operative
Total analgesic use postoperatively | from end of procedure to 24 hours post procedure
  analgesic use in the post operative period will be calculated in morphine equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Paul Miller, JDMD, Study Chair — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT07101250/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT07101250/ICF_001.pdf